CLINICAL TRIAL: NCT06879171
Title: Radiographic and Histomorphometric Assessment for Alveolar Ridge Preservation Using Autogenous Tooth Graft From Extracted Tooth Combined With Simvastatin 1:1 Versus Autogenous Tooth Graft: A Randomized Clinical Trial (RCT)
Brief Title: Radiographic and Histomorphometric Assessment for Alveolar Ridge Preservation Using Autogenous Tooth Graft From Extracted Tooth Combined With Simvastatin 1:1 Versus Autogenous Tooth Graft
Acronym: ARP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Mohamed Abd Elwhab, dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alveolar Ridge Preservation AT
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-03

CONDITIONS: Alveolar Ridge Preservation; Horizontal Alveolar Bone Loss; Vertical Alveolar Bone Loss; Delayed Implant; Autogenous Tooth Graft
Keywords: autogenous tooth graft; simvastatin; delayed implant; alveolar ridge preservation

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial (RCT) with parallel group ,two arms, with 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: Study participants will be blinded and each patient will be given a code by the researcher (N.M). Blinding of the investigator (N.M) isn't applicable. Biostatistician will be blinded. Participants' identity and their corresponding study group will be concealed by assigning an identification number to all laboratory specimens, data files and reports for the transfer data to and from assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- autogenous tooth graft combined with simvastatin 1:1 (Experimental): Test group : autogenous tooth graft from the extracted tooth combined with simvastatin drug with a ratio 1:1
  Interventions: Procedure: Alveolar ridge preservation
- Autogenous tooth graft (Active Comparator): Control group : Autogenous tooth graft
  Interventions: Procedure: Alveolar ridge preservation

INTERVENTIONS:
Procedure: Alveolar ridge preservation — Grafting of the socket with Autogenous tooth graft mixed with simvastatin immediately after tooth extraction
  Arms: autogenous tooth graft combined with simvastatin 1:1
Procedure: Alveolar ridge preservation — Grafting the socket with Autogenous tooth graft immediately after tooth extraction
  Arms: Autogenous tooth graft

SUMMARY:
This study will be held to overcome the previous limitations related to bone loss after teeth extraction by taking advantages from both Autogenous tooth graft and Simvastatin which will offer a promising synergistic approach for reducing alveolar ridge resorption, enhance bone regeneration and ensuring implant site development for future implant placement. This combination will address the gap in knowledge and offering a novel approach in alveolar ridge preservation. The Autogenous tooth graft will provide a scaffold and growth factor source for bone regeneration while Simvastatin will promotes osteogensis and angiogensis at graft site. So The goal of the present trial aims to evaluate the first-time application of Autogenous tooth graft from extracted tooth combined with Simvastatin with a ratio 1:1(test group) versus Autogenous tooth graft alone (control group) at an extraction socket of non molar single rooted teeth for alveolar ridge preservation and implant site development prior to implant placement.

The participants will be divided into two groups:

Intervention Group will receive Autogenous tooth graft combine with Simvastatin with a ratio 1:1 Control Group will receive Autogenous tooth graft. with follow up period 4 months.

DETAILED DESCRIPTION:
Alveolar ridge resorption following tooth extraction is one of the greatest challenges in dentistry, especially for patients seeking dental implants. The alveolar ridge undergoes significant decrease in bone dimensions which will complicate the implant placement and thus necessitate additional grafting procedures to compensate the bone loss. Bone height decreases progressively by 25% during the first year after tooth loss, with a total of 4 mm of height lost during this first year post-extraction.

So various grafting materials such as Autogenous bone grafts, bone substitutes and allografts, are adopted to overcome this challenge and preserve the alveolar ridge. Autogenous grafts are always the gold standard and the benchmark of all graft types because of Its osteoinductive, osteoconductive, and osteogenic. However, secondary surgical sites, pain, high rates of donor site morbidity, and limited supply of graft material are the main disadvantages of autogenous graft.

Among these also, Autogenous tooth graft the promising solution due to its biocompatibility, osteogenic properties and nature compositions that mimics the structure and function of lost bone.

Autogenous tooth graft a type of autogenous grafting technique that utilizes the extracted tooth/teeth of the same individual for the preparation of the graft material. A relatively new and innovative bone graft material with all the advantages of autogenous bone owing to its very similar components to bone and can be very useful in a multitude of clinical situations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with badly broken, non-restorable, or periodontally hopeless non molar single rooted teeth.
* Age from 20-45 years old(6,13). No sex predilection.
* Medically free from any medical condition that would interfere with bone healing.
* Patients with status classification (ASA I & II) with adequate oral hygiene condition.
* Alveolar sockets free from any preexisting periapical pathology based on intraoral periapical or panoramic radiograph.

Exclusion Criteria:

* Patients with any medical condition that contraindicated the procedure and general contraindications for Implant Surgery(6,13)
* Patients who are allergic to Simvastatin drug.(6)
* Presence of active infection around the tooth or remaining root.
* Psychological reasons that might affect the procedure or the subsequent follow up visits.
* Heavy smokers
* Immunosuppressed or Immunocompromised.(13)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone width | 4 months after grafting
  Pre- and Post-ARP CBCT Scans immediately and 4 months after grafting The scans will be compared using predetermined reference points to assess the bone width changes.

SECONDARY OUTCOMES:
vertical bone height | 4 months after grafting
  Pre- and Post-ARP CBCT Scans will be taken immediately and after 4 months of grafting.
  The scans will be compared using predetermined reference points to assess bone height changes.
percentage of newly formed bone | 4 months
  histomorphometrical analysis of the percentage of newly formed bone through decalcified bone sections with H&E stain using image analyzer computer Software.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Galal professor, phd holder, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Janjua OS, Qureshi SM, Shaikh MS, Alnazzawi A, Rodriguez-Lozano FJ, Pecci-Lloret MP, Zafar MS. Autogenous Tooth Bone Grafts for Repair and Regeneration of Maxillofacial Defects: A Narrative Review. Int J Environ Res Public Health. 2022 Mar 20;19(6):3690. doi: 10.3390/ijerph19063690. PMID 35329377
- [Background] Beca-Campoy T, Sanchez-Labrador L, Blanco-Antona LA, Cortes-Breton Brinkmann J, Martinez-Gonzalez JM. Alveolar ridge preservation with autogenous tooth graft: A histomorphometric analysis of 36 consecutive procedures. Ann Anat. 2025 Feb;258:152375. doi: 10.1016/j.aanat.2025.152375. Epub 2025 Jan 6. PMID 39778754
- [Background] Zhang S, Li X, Qi Y, Ma X, Qiao S, Cai H, Zhao BC, Jiang HB, Lee ES. Comparison of Autogenous Tooth Materials and Other Bone Grafts. Tissue Eng Regen Med. 2021 Jun;18(3):327-341. doi: 10.1007/s13770-021-00333-4. Epub 2021 Apr 30. PMID 33929713
- See also: https://pmc.ncbi.nlm.nih.gov/articles/PMC5822533/ — https://pmc.ncbi.nlm.nih.gov/articles/PMC8955500/